CLINICAL TRIAL: NCT06241183
Title: Comparing Intravenous Famotidine and Oral Antacids in the Treatment of Dyspepsia in the Emergency Department
Brief Title: Famotidine and Antacids for Treatment of Dyspepsia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Singer, Professor and Interim Chair of the Department of Emergency Medicine, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2023-00188
Record Dates: First submitted 2024-01-16; First posted 2024-02-05 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Dyspepsia; GERD; Acid Reflux
Keywords: dyspepsia; GERD; Acid Reflux; H2 receptor antagonist; antacid; Maalox; Mylanta; Famotidine
MeSH Terms: conditions — Dyspepsia; Gastroesophageal Reflux | interventions — Histamine H2 Antagonists; aluminum hydroxide, magnesium hydroxide, drug combination; aluminum hydroxide, magnesium hydroxide, simethicone drug combination; Antacids

STUDY DESIGN:
Intervention Model Description: Subjects are divided into two groups and randomly assigned to receive either study drug.
Who Masked: Outcomes Assessor
Masking Description: The research team member assessing verbal pain score will be blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Famotidine (Active Comparator): Patients in this group will receive 20 mg of intravenous famotidine.
  Interventions: Drug: Intravenous Famotidine
- Oral Maalox (Active Comparator): Patients in the group will receive 30 ml of oral Maalox/ Mylanta.
  Interventions: Drug: Oral Maalox/ Mylanta

INTERVENTIONS:
Drug: Intravenous Famotidine — Patients in this group will receive 20mg IV Famotidine.
  Other Names: H2 Receptor Antagonist
  Arms: Intravenous Famotidine
Drug: Oral Maalox/ Mylanta — Patients in this group will receive 30 ml Maalox/ Mylanta.
  Other Names: Antacid
  Arms: Oral Maalox

SUMMARY:
The aim of this study is to compare intravenous famotidine, an H2 receptor antagonist, and Maalox/ Mylanta, an oral antacid, in treatment of dyspepsia in the emergency department. The goal of this study is to reduce patients' pain based on the verbal numerical pain scale. The anticipated outcome is for pain levels in both groups to decrease. It is expected that antacids will improve symptoms more quickly and to a greater degree within an hour of taking medication based on the results of similar studies.

DETAILED DESCRIPTION:
This study will be conducted in the Emergency Department at Stony Brook University Hospital. Investigators intend to enroll approximately 80 patients who present to the emergency department with dyspepsia symptoms. The patients will be randomized to one of two groups: one group will receive 20 mg of intravenous famotidine and the other will receive 30 ml of oral Maalox/ Mylanta. The verbal numeric pain score (VNP) will be used to measure pain at 0 minutes, 15 minutes, 30 minutes, 45 minutes, and 60 minutes after administration of the study drug. Pain severity assessments will be performed by an investigator blinded to study treatment. Data will also be collected regarding demographic, clinical information, patient satisfaction and the need for rescue medications in each of the two study groups at the end of the 60-minute study period. At the end of the study period, the patients may be treated with additional analgesia at the discretion of their ED provider.

ELIGIBILITY:
Inclusion Criteria:

1. Subject Age ≥ 18 years of age
2. Patient diagnosed with dyspepsia
3. Present at the ED with upper abdominal pain score of at least 3

Exclusion Criteria:

1. Hypersensitivity to an ingredient in Maalox/ Mylanta or Famotidine
2. Moderate to Severe Renal Insufficiency (precaution)
3. Kidney Failure
4. Pregnant or Nursing
5. Verbal pain score less than 3
6. Inability to tolerate oral medications
7. Bowel Obstruction
8. Proton pump inhibitor within 2 hours of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Verbal Numerical Pain Score | at 1 hour
  Patients will be asked to rate their pain on a scale of 0 to 10 with 0 indicating no pain and 10 indicating the worst pain imaginable every 15 minutes for 60 minutes.

SECONDARY OUTCOMES:
Need for Rescue Medications | at 1 hour
  Investigators will assess frequency of need for rescue medications between groups.
Satisfaction with Assigned Medication | at 1 hour
  Investigators will gather data regarding patient satisfaction with their assigned treatment using a 5 item likert scale from very dissatisfied (1), dissatisfied (2) neither satisfied nor dissatisfied (3), satisfied (4) and very satisfied (5). The outcome will be measured as the percentages of patients choosing very satisfied or satisfied with their assigned medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No